CLINICAL TRIAL: NCT05516082
Title: Clinical Evaluation of Two Daily Disposable Lenses in Sphere Design
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: EX-MKTG-141
Record Dates: First submitted 2022-08-23; First posted 2022-08-25 (Actual); Results first posted 2023-11-28 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2022-10

CONDITIONS: Ametropia
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Intervention Model Description: All participants received Lens A and then Lens B in fixed-sequence order.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Lens A (Experimental): All participants wore Lens A for 15 minutes (Period 1)
  Interventions: Device: Lens A
- Lens B (Experimental): All participants wore Lens B for 15 minutes (Period 2)
  Interventions: Device: Lens B

INTERVENTIONS:
Device: Lens A — DDH contact lens for 15 minutes
  Arms: Lens A
Device: Lens B — DDSH contact lens for 15 minutes
  Arms: Lens B

SUMMARY:
This was a single-blind, interventional, prospective, direct refit, bilateral wear, fixed-sequence crossover study.

DETAILED DESCRIPTION:
The aim of this study was to evaluate the visual performance and subjective experiences of daily disposable hydrogel lens (DDH) when compared to daily disposable silicone hydrogel lens (DDSH) after 15 minutes of daily wear each.

ELIGIBILITY:
Inclusion Criteria:

* Is at least 18 years of age and has full legal capacity to volunteer.
* Has read and signed an information consent letter.
* Self-reports having a full eye examination in the previous two years.
* Anticipates being able to wear the study lenses for the required time of the study.
* Is willing and able to follow instructions and maintain the appointment schedule.
* Has refractive astigmatism no higher than -0.75 DC.
* Can be fit with the available lens parameters (sphere +8.00 to -10.00D).
* Can achieve binocular distance vision of at least 20/30 Snellen (logMAR 0.18) with the study contact lenses.

Exclusion Criteria:

* Is participating in any concurrent clinical or research study.
* Has any known active ocular disease and/or infection that contraindicates contact lens wear.
* Has a systemic condition that in the opinion of the investigator may affect a study outcome variable.
* Is using any systemic or topical medications that in the opinion of the investigator may affect contact lens wear or a study outcome variable.
* Has known sensitivity to the diagnostic sodium fluorescein used in the study.
* Self-reports as pregnant, lactating or planning a pregnancy at the time of enrolment.
* Has undergone refractive error surgery or intraocular surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2022-08-08 (Actual); Primary Completion 2022-10-12 (Actual); Study Completion 2022-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rubén V Guerrero, MSc., FIACLE, Principal Investigator — Dr. Ruben Velazquez Private Practice
Locations (1):
- Dr. Ruben Velazquez Private Practice, Mexico City, Mexico

RESULTS

PARTICIPANT FLOW:
Groups:
- Lens A (DDH Contact Lens): All participants wore Lens A for 15 minutes (Period 1)
- Lens B (DDSH Contact Lens): All participants wore Lens B for 15 minutes (Period 2)
Period: Period 1: Lens A, 15 Minutes
Arm/Group | Lens A (DDH Contact Lens) | Lens B (DDSH Contact Lens)
Started | 41 | 0 (All participants received Lens A in Period 1.)
Completed | 41 | 0
Not Completed | 0 | 0
Period: Period 2: Lens B, 15 Minutes
Arm/Group | Lens A (DDH Contact Lens) | Lens B (DDSH Contact Lens)
Started | 0 (All participants received Lens B in Period 2.) | 41
Completed | 0 | 41
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Includes all study participants.
Arm/Group | All Study Participants
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.6 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Lens Fit Acceptance
Description: Measured on a scale of 0-4 (0 = Should not be worn, 1 = Borderline but unacceptable, 2 = Min. acceptable, early review, 3 = Not perfect but OK to dispense, 4 = Perfect) as assessed by an investigator.
Time Frame: 15 minutes
Population: All participants wore Lens A and Lens B in sequential order.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Lens A: Participants that received Lens A.
- Lens B: Participants that received Lens B.
Arm/Group | Lens A | Lens B
Number analyzed (Participants) | 41 | 41
score on a scale | 3.51 (0.9) | 3.68 (0.7)

ADVERSE EVENTS:
Time Frame: From dispense up to 15 minutes on each lens type
Arm/Group | Lens A | Lens B
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/41
Other Adverse Events (participants affected / at risk) | 0/41 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-18): https://cdn.clinicaltrials.gov/large-docs/82/NCT05516082/Prot_SAP_000.pdf